CLINICAL TRIAL: NCT01664858
Title: Clinical Evaluation of Magnetic Resonance Imaging in Coronary Heart Disease - 2 (CE-MARC2)
Brief Title: Clinical Evaluation of Magnetic Resonance Imaging in Coronary Heart Disease-2
Acronym: CE-MARC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Leicester (Other); University of Glasgow (Other); British Heart Foundation (Other)
Responsible Party: Principal Investigator, Professor JP Greenwood, Professor of Cardiology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SP/12/1/29062
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-05

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Ischaemic Heart Disease; Angina; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3T CMR-guided management (Active Comparator): Patient to be managed according to the results of 3T CMR imaging
  Interventions: Other: 3T CMR; Other: X-Ray coronary angiography
- SPECT-guided management (Active Comparator): Patients to be managed according to the results of SPECT
  Interventions: Other: SPECT; Other: X-Ray coronary angiography
- NICE-guidelines based management (Active Comparator): Patients will be receive NICE-guidelines based management and will receive the imaging strategy specified by NICE according to their pre-test likelihood of having CHD.
  10-29% - CT calcium score +/- CT coronary angiography; 30-60% - SPECT; 61-90% - X-Ray coronary angiography
  Interventions: Other: SPECT; Other: CT calcium score; Other: CT coronary angiography; Other: X-Ray coronary angiography

INTERVENTIONS:
Other: 3T CMR — 3Tesla Cardiac Magnetic Resonance Imaging
  Arms: 3T CMR-guided management
Other: SPECT — SPECT: Single Photon Emission Computed Tomography
  Arms: NICE-guidelines based management; SPECT-guided management
Other: CT calcium score — CT calcium score
  Arms: NICE-guidelines based management
Other: CT coronary angiography — CT coronary angiography
  Arms: NICE-guidelines based management
Other: X-Ray coronary angiography — X-Ray coronary angiography

SUMMARY:
CE-MARC 2 is a randomised controlled trial to determine diagnosis and patient management in patients presenting to outpatient clinics with suspected stable angina. Cardiac Magnetic Resonance Imaging (at 3Tesla) will be evaluated prospectively against current best clinical practice (defined by international guidelines). The study hypothesis is that 3Tesla CMR-guided management of patients with suspected stable angina is superior to current clinical practice based on 1) the principles of the National Institutes for Clinical Excellence (NICE) CG95 guidelines (2010); 2) SPECT AHA appropriateness criteria, in terms of avoiding study-defined unnecessary invasive coronary angiography.

DETAILED DESCRIPTION:
The study is a randomized controlled trial of non-invasive imaging to determine diagnosis and management of patients presenting with suspected stable angina. Despite the widespread availability of non-invasive imaging and guideline-enshrined use of optimal medical therapy (OMT), patients with suspected coronary heart disease (CHD) often end up having invasive coronary angiography early in their disease course. Currently >50% of elective invasive coronary angiograms performed in the UK and US do not lead on to a revascularisation procedure (data from 2008-09 UK Hospital Episode Statistics; American College of Cardiology National Cardiovascular Data Registry (Patel MR, et al., N Engl J Med 2010;362:886-95)). The UK NICE guidelines for the management of chest pain of recent onset (CG95; 2010) could increase this proportion even further. This is inefficient for patients and also of healthcare resources.

More widespread use of non-invasive functional imaging could reduce the rates of unnecessary angiography. We have shown in the CE-MARC study (Lancet 2012) that cardiovascular magnetic resonance (CMR) at 1.5Tesla has a higher diagnostic accuracy for the detection of CHD than single-photon emission computed tomography (SPECT). CE-MARC 2 will be a three-way randomised controlled trial of patient management in 1200 patients with known or suspected CHD, comparing 3Tesla CMR to SPECT-guided care or NICE guidelines-based management. The primary endpoint will be the reduction of unnecessary invasive angiography (defined by invasive FFR) at 12 months - identified by our expert patients as an important 'patient focused' clinical outcome measure. The secondary objectives will include: 1) assessment of safety of a CMR-guided management strategy 2) cost effectiveness analysis of these strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥30yrs
* Patient has suspected stable angina (CHD) that requires further investigation
* Has a defined risk of 10-90% (according to NICE guidelines CG95; 2010)
* Suitable for revascularisation if required
* Given informed written consent

Exclusion Criteria:

* Non-anginal chest pain
* Clinically unstable
* Previous MI or biomarker positive ACS
* Previous revascularisation with coronary artery bypass surgery or PCI
* Contraindication to CMR imaging (pacemaker, intra-orbital debris, intra-auricular implants, intracranial clips, severe claustrophobia)
* Contraindication to adenosine infusion (regular adenosine antagonist medication, significant reversible airways disease, second or third degree atrio-ventricular heart block, sino-atrial disease)
* Known adverse reaction to Adenosine or Gadolinium contrast agent
* Obesity (where body girth exceeds scanner diameter)
* Pregnancy or breast feeding
* Inability to give informed consent
* Known chronic renal failure (eGFR <30mL/min/1.73m2)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Greenwood, PhD, Principal Investigator — University of Leeds
Locations (6):
- United Kingdom (6):
  - Glenfield Hospital, Leicester, Leicestershire
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - University Hospitals Bristol NHS FT, Bristol
  - Golden Jubilee National Hospital, Glasgow
  - St Georges Healthcare NHS Trust, London
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ripley DP, Brown JM, Everett CC, Bijsterveld P, Walker S, Sculpher M, McCann GP, Berry C, Plein S, Greenwood JP. Rationale and design of the Clinical Evaluation of Magnetic Resonance Imaging in Coronary heart disease 2 trial (CE-MARC 2): a prospective, multicenter, randomized trial of diagnostic strategies in suspected coronary heart disease. Am Heart J. 2015 Jan;169(1):17-24.e1. doi: 10.1016/j.ahj.2014.10.008. Epub 2014 Oct 22. PMID 25497243
- [Result] Greenwood JP, Ripley DP, Berry C, McCann GP, Plein S, Bucciarelli-Ducci C, Dall'Armellina E, Prasad A, Bijsterveld P, Foley JR, Mangion K, Sculpher M, Walker S, Everett CC, Cairns DA, Sharples LD, Brown JM; CE-MARC 2 Investigators. Effect of Care Guided by Cardiovascular Magnetic Resonance, Myocardial Perfusion Scintigraphy, or NICE Guidelines on Subsequent Unnecessary Angiography Rates: The CE-MARC 2 Randomized Clinical Trial. JAMA. 2016 Sep 13;316(10):1051-60. doi: 10.1001/jama.2016.12680. PMID 27570866
- [Derived] Everett CC, Berry C, McCann GP, Fernandez C, Reynolds C, Bucciarelli-Ducci C, Dall'Armellina E, Prasad A, Foley JR, Mangion K, Bijsterveld P, Brown J, Stocken D, Walker S, Sculpher M, Plein S, Greenwood JP. Randomised trial of stable chest pain investigation: 3-year clinical and quality of life results from CE-MARC 2. Open Heart. 2023 May;10(1):e002221. doi: 10.1136/openhrt-2022-002221. PMID 37130657
- [Derived] Corcoran D, Young R, Adlam D, McConnachie A, Mangion K, Ripley D, Cairns D, Brown J, Bucciarelli-Ducci C, Baumbach A, Kharbanda R, Oldroyd KG, McCann GP, Greenwood JP, Berry C. Coronary microvascular dysfunction in patients with stable coronary artery disease: The CE-MARC 2 coronary physiology sub-study. Int J Cardiol. 2018 Sep 1;266:7-14. doi: 10.1016/j.ijcard.2018.04.061. Epub 2018 Apr 19. PMID 29716756

RESULTS

PARTICIPANT FLOW:
Groups:
- NICE-guidelines Based Management: Patients will be receive NICE-guidelines based management and will receive the imaging strategy specified by NICE according to their pre-test likelihood of having CHD.
  10-29% - CT calcium score +/- CT coronary angiography; 30-60% - SPECT; 61-90% - X-Ray coronary angiography
  SPECT: SPECT: Single Photon Emission Computed Tomography
  CT calcium score: CT calcium score
  CT coronary angiography: CT coronary angiography
  X-Ray coronary angiography: X-Ray coronary angiography
Period: Overall Study
Arm/Group | 3T CMR-guided Management | SPECT-guided Management | NICE-guidelines Based Management
Started | 481 | 481 | 240
Completed | 467 | 468 | 234
Not Completed | 14 | 13 | 6

BASELINE CHARACTERISTICS:
Groups:
- 3T CMR-guided Management: Patient to be managed according to the results of 3T CMR imaging
  3T CMR: 3Tesla Cardiac Magnetic Resonance Imaging
  X-Ray coronary angiography: X-Ray coronary angiography
  Patients with suspected angina pectoris were eligible if they were 30 years or older, had a CHD pretest likelihood of 10% to 90%, and suitable for revascularization. Exclusion criteria included nonanginal chest pain, a normal MPS or cardiac computed tomography (CCT) result within the previous 2 years, being clinically unstable, previous myocardial infarction, previous coronary revascularization, and contraindication to any study noninvasive imaging test .
- SPECT-guided Management: Patients to be managed according to the results of SPECT
  SPECT: SPECT: Single Photon Emission Computed Tomography
  X-Ray coronary angiography: X-Ray coronary angiography
  Patients with suspected angina pectoris were eligible if they were 30 years or older, had a CHD pretest likelihood of 10% to 90%, and suitable for revascularization. Exclusion criteria included nonanginal chest pain, a normal MPS or cardiac computed tomography (CCT) result within the previous 2 years, being clinically unstable, previous myocardial infarction, previous coronary revascularization, and contraindication to any study noninvasive imaging test .
- NICE-guidelines Based Management: Patients will be receive NICE-guidelines based management and will receive the imaging strategy specified by NICE according to their pre-test likelihood of having CHD.
  10-29% - CT calcium score +/- CT coronary angiography; 30-60% - SPECT; 61-90% - X-Ray coronary angiography
  SPECT: SPECT: Single Photon Emission Computed Tomography
  CT calcium score: CT calcium score
  Patients with suspected angina pectoris were eligible if they were 30 years or older, had a CHD pretest likelihood of 10% to 90%, and suitable for revascularization. Exclusion criteria included nonanginal chest pain, a normal MPS or cardiac computed tomography (CCT) result within the previous 2 years, being clinically unstable, previous myocardial infarction, previous coronary revascularization, and contraindication to any study noninvasive imaging test .
  CT coronary angiography: CT coronary angiography
  X-Ray coronary angiography: X-Ray coronary angiography
- Total: Total of all reporting groups
Arm/Group | 3T CMR-guided Management | SPECT-guided Management | NICE-guidelines Based Management | Total
Number analyzed (Participants) | 481 | 481 | 240 | 1202
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.10) | 55.9 (8.87) | 56.5 (9.21) | 56.3 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227 | 225 | 112 | 564
  Male | 254 | 256 | 128 | 638

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unnecessary Invasive Coronary Angiography
Description: * A negative FFR and positive non-invasive test (either 3T CMR or SPECT/CCT)
  * A negative FFR in a high pre-test risk (61-90%) patient that proceeds directly to invasive angiography in the NICE guidelines-based strategy arm
  * A negative FFR and a negative non-invasive test (either 3T CMR or SPECT/CCT) (i.e. a True Negative strategy result in which the imaging result was 'not believed' by the treating cardiologist)
  * An inconclusive non-invasive test result (either 3T CMR or SPECT/CCT) in which angiography had to be performed to make the diagnosis
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 3T CMR-guided Management | SPECT-guided Management | NICE-guidelines Based Management
Number analyzed (Participants) | 481 | 481 | 240
Participants | 36 | 34 | 69

2. Secondary Outcome: Major Adverse Cardiovascular Event (MACE)
Description: MACE is defined as one of the following:
  * Death due to cardiovascular cause (including type 3 MI) †
  * Myocardial infarction†
  * Unplanned revascularisation
  * Hospital admission for cardiovascular cause [ACS Troponin -ve, spontaneous myocardial infarction (Type 1)†, Myocardial infarction secondary to ischaemic imbalance (Type 2) †, Myocardial Infarction related to stent thrombosis (Type 4b) †, Arrhythmia, Stroke, Heart failure]. † As defined by the third universal definition of myocardial infarction.
Time Frame: at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 3T CMR-guided Management | SPECT-guided Management | NICE-guidelines Based Management
Number analyzed (Participants) | 481 | 481 | 240
Participants | 20 | 17 | 4

3. Secondary Outcome: Positive Angiogram (by FFR) Rate for Each Strategy.
Description: The Positive Angiogram rate will be determined from the proportion of patients in the relevant population who undergo an angiogram within 12 months of randomisation which yields a positive finding by FFR (or QCA where no FFR reading is undertaken)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 3T CMR-guided Management | SPECT-guided Management | NICE-guidelines Based Management
Number analyzed (Participants) | 481 | 481 | 240
Participants | 47 | 42 | 29

4. Secondary Outcome: Cost Effectiveness Analysis
Description: To assess the long term cost-effectiveness of the alternate diagnostic testing strategies, information from the trial will be used to update the economic model developed as part of the original CE-MARC trial. The model will use information from the trial, including on resource use, costs, HRQoL and other clinical outcomes (e.g. on unnecessary tests and MACE events), together with epidemiological, clinical and economic data from other sources to calculate costs and quality-adjusted life-years (QALYs) for patients. The economic analysis will use methods consistent with those recommended by the National Institute for Health and Clinical Excellence (NICE). Given the potential difference between diagnostic strategies in terms of mortality, the modelling will adopt a lifetime time horizon to capture any difference.
Time Frame: 3 years
Reporting Status: Not Posted

5. Secondary Outcome: Health-related Quality-of-life Measures (SAQ-UK; SF12; EQ-5D)
Description: Health-related quality-of-life (HRQoL) will be measured at baseline (in clinic), 6 months, 12 months, 2yrs and 3yrs (by post), using the following validated questionnaires:
  * Seattle Angina Questionnaire (SAQ) - UK version
  * SF12v2
  * EuroQol (EQ-5D)
Time Frame: 3 years
Reporting Status: Not Posted

6. Secondary Outcome: Complications
Description: Complications - investigational or procedural related only. All complications from all study procedures/investigations will be recorded and reported if they result in an extended length of stay or specific treatment.
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Description: MACEs: cardiovascular death, myocardial infarction, unplanned coronary revascularization, and hospital admission for cardiovascular cause.
Arm/Group | 3T CMR-guided Management | SPECT-guided Management | NICE-guidelines Based Management
Serious Adverse Events (participants affected / at risk) | 15/481 | 15/481 | 6/240
Other Adverse Events (participants affected / at risk) | 6/481 | 0/481 | 2/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3T CMR-guided Management (N=481) | SPECT-guided Management (N=481) | NICE-guidelines Based Management (N=240)
Major Adverse Cardiovascular Event (Cardiac disorders) | 15 (20) | 15 (17) | 6 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3T CMR-guided Management (N=481) | SPECT-guided Management (N=481) | NICE-guidelines Based Management (N=240)
Expected Test Complication (Investigations) | 6 (6) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No